CLINICAL TRIAL: NCT01458613
Title: Biomarker for Maroteaux-Lamy Disease: BioMaroteaux-Lamy AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Maroteaux-Lamy Disease (BioMaroteaux)
Acronym: BioMaroteaux
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BMAL 06-2018
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Lysosomal Storage Disease; Lung Diseases; Obstructive Sleep Apnoea; Macroglossia; Eye Abnormalities
Keywords: Maroteaux-Lamy Disease; Biomarker
MeSH Terms: conditions — Lysosomal Storage Diseases; Lung Diseases; Sleep Apnea, Obstructive; Macroglossia; Eye Abnormalities; Mucopolysaccharidosis VI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of mass-spectometry 10 ml EDTA blood or a dry blood spot filter card are taken. To proof the correct Maroteaux-Lamy diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Maroteaux-Lamy will be done as routine diagnostic.
  The analyses will be done at the:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Maroteaux-Lamy disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Maroteaux-Lamy disease from blood

DETAILED DESCRIPTION:
Maroteaux-Lamy disease (MPS VI) is a lysosomal storage disease inherited in an autosomal recessive pattern. The responsible mutations lie in ARSB (5q11-q13), the gene that encodes the enzyme arylsulfatase B. The phenotype results from defective dermatan sulfate break-down with lysosomal accumulation. This accumulation of glycosaminoglycans is responsible for the widespread signs and symptoms found in this disease. Bone destruction in shoulders, hips and skull is often seen by the second decade of life and may become evident later in the knees and spine. Early growth may be normal but eventually slows resulting in short stature. Dysplasia of bones comprising these joints leads to stiffness and restricted movement. The face is dysmorphic with coarse features. Bone dysplasia and facial dysmorphism may be seen at birth.

Myelopathy and even tetraplegia can result from vertebral compression. Intelligence is often normal although more severely affected individuals may have some cognitive defects due to impaired vision and hearing. Hepatosplenomegaly is common and compromised respiratory function can result in reduced physical stamina. The tongue is usually enlarged. Accumulation of dermatan sulfate in heart valves may produce insufficiency or restriction of outflow. A diagnosis of Maroteaux-Lamy disease can be confirmed by screening for the common genetic mutations or measuring the level of the arylsulfatase B enzyme activity in a blood sample -- a test that has 100 percent accuracy. Once Maroteaux-Lamy disease is diagnosed, testing of all family members and consultation with a professional geneticist is recommended. Carriers are most reliably identified via genetic mutation analysis.

New methods, like mass-spectrometry give a good chance to characterize in the blood (plasma) of affected patents specific metabolic alterations that allow to diagnose in the future the disease earlier, with a higher sensitivity and specificity. Therefore it is the goal of the study to develop new biochemical markers from the plasma of the affected patients helping to benefit the patient by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients older than 12 months
* The patient has a diagnosis of Maroteaux-Lamy disease

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures
* Patients younger than 12 months
* The patient has no diagnosis of Maroteaux-Lamy disease

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Maroteaux-Lamy disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Maroteaux-Lamy disease from blood (plasma) | 24 month
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided